CLINICAL TRIAL: NCT00381706
Title: Randomized Phase II Study of ECF-C, IC-C, or FOLFOX-C in Metastatic Esophageal and GE Junction Cancer
Brief Title: Combination Chemotherapy and Cetuximab in Treating Patients With Metastatic Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Bristol-Myers Squibb (Industry); Sanofi (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80403; ECOG-E1206; CDR0000505535 (Other: Physician Data Query); NCI-2009-00492 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Cancer
Keywords: squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus; stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cetuximab; Epirubicin; Fluorouracil; Cisplatin; Irinotecan; Folfox protocol; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (ECF + cetuximab) (Experimental): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab IV on days 1, 8 and 15. Patients receive epirubicin 50 mg/m^2 IV after cetuximab on day 1 followed by cisplatin 60 mg/m^2 IV over 60 minutes. On days 1-21, patients receive 5-fluorouracil 200 mg/m^2/day continuous IV infusion. Treatment repeats every 21 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: ECF
- Arm B (IC + cetuximab) (Experimental): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab on days 1, 8 and 15. Patients receive cisplatin 30 mg/m^2 IV over 30 minutes on days 1 and 8 after cetuximab. Patients also receive irinotecan 65 mg/m^2 IV over 90 minutes on days 1 and 8 after receiving cisplatin.Treatment repeats every 21 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: IC
- ARM C (FOLFOX + cetuximab) (Experimental): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab on days 1 and 8. On Day 1, patients also receive oxaliplatin 85 mg/m^2 IV over 120 minutes and leucovorin 400 mg/m^2 IV over 120 minutes either concurrently with oxaliplatin via a separate infusion line or post oxaliplatin administration. Following leucovorin, patients will receive 5-fluorouracil 400 mg/m^2 IV bolus injection, then 5-fluorouracil 2400 mg/m^2 IV infusion over 46-48 hours. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: FOLFOX

INTERVENTIONS:
Biological: cetuximab — given IV
  Other Names: C225
Drug: ECF — epirubicin and 5-fluorouracil given IV
  Other Names: Ellence (epirubicin) and 5-fluorouracil (5-FU)
  Arms: Arm A (ECF + cetuximab)
Drug: IC — cisplatin and irinotecan given IV
  Other Names: Platinol-AQ (cisplatin), CPT-11 (irinotecan)
  Arms: Arm B (IC + cetuximab)
Drug: FOLFOX — oxaliplatin , leucovorin and 5-fluorouracil IV
  Other Names: Eloxatin (oxaliplatin), folinic acid (leucovorin), and 5-fluorouracil (5-FU)
  Arms: ARM C (FOLFOX + cetuximab)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one chemotherapy drug (combination chemotherapy) together with cetuximab may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying three different combination chemotherapy regimens to compare how well they work when given together with cetuximab in treating patients with metastatic esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, multicenter study. Patients are stratified according to histology (squamous cell carcinoma vs adenocarcinoma) and Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 vs 2). Patients are randomized to 1 of 3 treatment arms. For more information please see the "Arms" section which includes a detailed description of the treatment regimens.

The primary objective of the study is evaluate the tumor response rate (RR) for each of the regimens in this trial and to select the most promising regimen based on RR for further testing in patients with metastatic esophageal or GE junction adenocarcinoma. The secondary objectives are:

1. To evaluate overall survival (OS) for each of the regimens in this trial in patients with metastatic esophageal or GE junction adenocarcinoma.
2. To evaluate progression-free survival (PFS) for each of the regimens in this trial in patients with metastatic esophageal or GE junction adenocarcinoma.
3. To evaluate time to treatment failure (TTF) for each of the regimens in this trial in patients with metastatic esophageal or GE junction adenocarcinoma.
4. To determine the type and severity of toxicities associated with each of these regimens in the multi-institutional phase II setting.
5. Quantitative immunohistochemistry results will be correlated with objective response rate, overall survival and time to progression.
6. To evaluate the cellular damage (apoptosis) as a result of oxaliplatin.
7. To determine if germline EGFR variants correlate with skin rash in patients treated with cetuximab.
8. To evaluate if a correlation exists between germline EGFR variants and tumor EFGR expression as measured by immunohistochemistry.

All subjects must be premedicated with diphenhydramine hydrochloride 50 mg IV (or a similar agent) prior to the first dose of cetuximab in an effort to minimize infusion and hypersensitivity reactions. Premedication is recommended prior to subsequent doses, but the dose of diphenhydramine (or similar agent) may be reduced at the investigator's discretion. More information is detailed in the protocol including a description of the premedication requirements. Patients were closely monitored for treatment-related adverse events. After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
1. Metastatic disease of the esophagus or gastroesophageal junction

   1. Histologic, cytologic or radiologic documentation of metastatic squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction. Radiologic, endoscopic, histologic or cytologic evidence of locally recurrent or locally residual (post-resection) disease is also permitted.
   2. For the purposes of this study, undifferentiated adenocarcinomas and adenosquamous tumors will be considered as adenocarcinomas. In addition, tumors involving the gastroesophageal junction will be defined by the Siewert classification.
   3. Patients with gastroesophageal junction tumors who are eligible:

      * AEG Type I: Adenocarcinoma of the distal esophagus which usually arises from an area with specialized intestinal metaplasia of the esophagus (eg, Barrett's esophagus, and may infiltrate the esophagogastric junction from above).
      * AEG Type II: True carcinoma of the cardia arising from the cardiac epithelium or short segments with intestinal metaplasia at the esophagogastric junction.
   4. Patients with gastroesophageal junction tumors who are NOT eligible:

      * AEG Type III: Subcardial gastric carcinoma which infiltrates the esophagogastric junction and distal esophagus from below.
2. Patients must have at least one paraffin block available (or at least 15 unstained slides for analysis of tumor EGFR status.

   1. Patients with a history of esophageal and GE junction carcinoma treated by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of greater than five years has elapsed between the primary surgery and the development of metastatic disease OR the primary cancer was stage I.
   2. Clinicians should consider biopsy of lesions to establish the diagnosis of metastatic esophageal or GE junction carcinoma if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
3. Patients with Measurable Disease - Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan.
4. Prior Treatment:

   1. No prior chemotherapy or radiotherapy. No prior therapy which specifically and directly targets the EGF(R) pathway.
   2. No prior allergic reaction to chimerized or murine monoclonal antibody therapy or documented presence of human anti-mouse antibodies (HAMA).
   3. Patients must have completed any major surgery ≥ 4 weeks or any minor surgery ≥ 2 weeks before registration. Patients must have fully recovered from the procedure. Insertion of a vascular access device is not considered major or minor surgery.
   4. No concurrent use of investigational agents is allowed while participating in this study.
5. Patient Characteristics:

   1. ECOG Performance Status of 0-2
   2. ≥ 18 years of age
   3. Patients must be documented to have a stable weight (or less than one pound weight loss) for at least one week prior to registration.
   4. Non-pregnant and not breast-feeding. The effects of cetuximab, cisplatin, epirubicin, fluorouracil, leucovorin, irinotecan, and oxaliplatin on a developing human fetus are not well-known. Because the risk of toxicity in nursing infants secondary to cetuximab, cisplatin, epirubicin, fluorouracil, irinotecan, and oxaliplatin treatment of the mother is unknown but may be harmful, breastfeeding must be discontinued.
6. No myocardial infarction < 6 months prior to registration or New York Heart Association classification III or IV.
7. No ≥ grade 2 diarrhea within 7 days prior to registration.
8. Patients may not concurrently have any of the following conditions:

   1. Known central nervous system metastases or carcinomatous meningitis
   2. Interstitial pneumonia or symptomatic interstitial fibrosis of the lung
   3. Seizure disorder or active neurological disease requiring anti-epileptic medication
   4. ≥ grade 2 peripheral neuropathy
9. No evidence of Gilbert's Syndrome - Patients with Gilbert's Syndrome may have a greater risk of irinotecan toxicity due to the abnormal glucuronidation of SN-38, the active metabolite of irinotecan. Evidence of Gilbert's Syndrome would include documentation of elevation of indirect bilirubin at any time in the patient's medical history.
10. Required Initial Laboratory Data:

    1. Granulocytes ≥ 1500/µl
    2. Platelet count ≥ 100,000/µl
    3. Creatinine ≤ 1.5 mg/dL
    4. AST (SGOT) ≤ 5.0 x Upper limits of normal
    5. Total bilirubin ≤ 1.5 mg/dL
    6. Albumin ≥ 2.5 grams/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-09-15 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2014-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Study Chair — Dana-Farber Cancer Institute
Locations (227):
- United States (227):
  - Norwalk Hospital, Norwalk, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Enzinger PC, Burtness BA, Niedzwiecki D, Ye X, Douglas K, Ilson DH, Villaflor VM, Cohen SJ, Mayer RJ, Venook A, Benson AB 3rd, Goldberg RM. CALGB 80403 (Alliance)/E1206: A Randomized Phase II Study of Three Chemotherapy Regimens Plus Cetuximab in Metastatic Esophageal and Gastroesophageal Junction Cancers. J Clin Oncol. 2016 Aug 10;34(23):2736-42. doi: 10.1200/JCO.2015.65.5092. Epub 2016 Jul 5. PMID 27382098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2006 and May 2009, 245 participants were enrolled and randomized.
Pre-assignment Details: Twenty three (23) participants had squamous cell carcinoma were excluded from the analysis.
Period: Overall Study
Arm/Group | Arm A (ECF + Cetuximab) | Arm B (IC + Cetuximab) | ARM C (FOLFOX + Cetuximab)
Started | 82 | 83 | 80
Completed | 75 | 81 | 79
Not Completed | 7 | 2 | 1
Not completed — Never treated | 7 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Adenocarcinoma (ECF + Cetuximab); Arm A: Squamous Cell Carcinoma (ECF + Cetuximab): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab IV on days 1, 8 and 15. Patients receive epirubicin 50 mg/m^2 IV after cetuximab on day 1 followed by cisplatin 60 mg/m^2 IV over 60 minutes. On days 1-21, patients receive 5-fluorouracil 200 mg/m^2/day continuous IV infusion. Treatment repeats every 21 days in the absence of disease progression and unacceptable toxicity.
- Arm B: Adenocarcinoma (IC + Cetuximab); Arm B: Squamous Cell Carcinoma (IC + Cetuximab): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab on days 1, 8 and 15. Patients receive cisplatin 30 mg/m^2 IV over 30 minutes on days 1 and 8 after cetuximab. Patients also receive irinotecan 65 mg/m^2 IV over 90 minutes on days 1 and 8 after receiving cisplatin.Treatment repeats every 21 days in the absence of disease progression and unacceptable toxicity.
- Arm C: Adenocarcinoma (FOLFOX + Cetuximab); Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab): Patients receive cetuximab 400 mg/m^2 IV over 120 minutes on day 1 of the first cycle, then 250 mg/m^2 IV over 60 minutes thereafter. Patients receive cetuximab on days 1 and 8. On Day 1, patients also receive oxaliplatin 85 mg/m^2 IV over 120 minutes and leucovorin 400 mg/m^2 IV over 120 minutes either concurrently with oxaliplatin via a separate infusion line or post oxaliplatin administration. Following leucovorin, patients will receive 5-fluorouracil 400 mg/m^2 IV bolus injection, then 5-fluorouracil 2400 mg/m^2 IV infusion over 46-48 hours. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab) | Arm A: Squamous Cell Carcinoma (ECF + Cetuximab) | Arm B: Squamous Cell Carcinoma (IC + Cetuximab) | Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab) | Total
Number analyzed (Participants) | 67 | 73 | 73 | 8 | 8 | 6 | 235
Age, Continuous [Median (Full Range); unit: years] | 57.7 [33 to 87] | 60.3 [34 to 81] | 59.2 [30 to 83] | 61.6 [52 to 84] | 61.8 [52 to 69] | 61.2 [50 to 76] | 59.3 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 5 | 2 | 3 | 1 | 32
  Male | 59 | 60 | 68 | 6 | 5 | 5 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 2 | 0 | 9
  White | 65 | 69 | 71 | 6 | 6 | 6 | 223
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 67 | 73 | 73 | 8 | 8 | 6 | 235

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial) in Patients With Measurable Esophageal or GE Junction Adenocarcinoma
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria. Overall tumor response is the total number of CR and PRs in participants with adenocarcinoma who have received at least one cycle of therapy.
Time Frame: Up to 2 years post-treatment
Population: 13 participants did not meet the protocol defined requirements to be evaluated for response (measurable adencarcinoma receiving at least 1 cycle of chemotherapy).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab)
Number analyzed (Participants) | 63 | 71 | 66
percentage of participants | 61 [48 to 72] | 45 [33 to 57] | 54 [42 to 66]

2. Secondary Outcome: Tumor Response Rate (Complete and Partial) in Patients With Squamous Cell Carcinoma
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria. Overall tumor response is the total number of CR and PRs in participants with squamous cell carcinoma who have received at least one cycle of therapy.
Time Frame: Up to 2 years post-treatment
Population: 4 participants did not meet the protocol defined requirements to be evaluated for response (measurable squamous cell carcinoma receiving at least 1 cycle of chemotherapy).
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Squamous Cell Carcinoma (ECF + Cetuximab) | Arm B: Squamous Cell Carcinoma (IC + Cetuximab) | Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab)
Number analyzed (Participants) | 6 | 8 | 5
percentage of participants | 67 | 13 | 60

3. Secondary Outcome: Overall Survival in Patients With Adenocarcinoma
Description: Overall survival (OS) was defined as the time from study entry to death of any cause. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 2 years post-treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab)
Number analyzed (Participants) | 67 | 73 | 73
months | 11.6 [8.1 to 13.4] | 8.6 [6.0 to 12.4] | 11.8 [8.8 to 13.9]

4. Secondary Outcome: Progression-free Survival in Patients With Adenocarcinoma
Description: Progression free survival (PFS) was defined as the time from study entry to progression or death of any cause. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 2 years post-treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab)
Number analyzed (Participants) | 67 | 73 | 73
months | 7.1 [4.5 to 8.4] | 4.9 [3.9 to 6.0] | 6.8 [5.4 to 8.1]

5. Secondary Outcome: Time to Treatment Failure in Patients With Adenocarcinoma
Description: Time to treatment failure (TTF) was measured from study entry until documented progression, death resulting from any cause, or end of protocol therapy because of unacceptable toxicity. The median TTF with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 2 years post-treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab)
Number analyzed (Participants) | 67 | 73 | 73
months | 5.6 [3.9 to 7.2] | 4.3 [3.6 to 5.5] | 6.7 [4.8 to 7.4]

ADVERSE EVENTS:
Arm/Group | Arm A: Adenocarcinoma (ECF + Cetuximab) | Arm B: Adenocarcinoma (IC + Cetuximab) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab) | Arm A: Squamous Cell Carcinoma (ECF + Cetuximab) | Arm B: Squamous Cell Carcinoma (IC + Cetuximab) | Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab)
Serious Adverse Events (participants affected / at risk) | 15/67 | 23/73 | 22/73 | 2/8 | 2/8 | 1/6
Other Adverse Events (participants affected / at risk) | 65/67 | 68/73 | 71/73 | 8/8 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Adenocarcinoma (ECF + Cetuximab) (N=67) | Arm B: Adenocarcinoma (IC + Cetuximab) (N=73) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab) (N=73) | Arm A: Squamous Cell Carcinoma (ECF + Cetuximab) (N=8) | Arm B: Squamous Cell Carcinoma (IC + Cetuximab) (N=8) | Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab) (N=6)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (11) | 12 (12) | 9 (10) | 2 (4) | 1 (1) | 1 (2)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 15 (17) | 8 (8) | 2 (3) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 8 (9) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (10) | 9 (9) | 1 (1) | 2 (2) | 1 (3)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (12) | 19 (21) | 15 (18) | 2 (4) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Sudden death (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jejunal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (4) | 3 (3) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 6 (7) | 8 (8) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 5 (5) | 4 (5) | 1 (2) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 10 (12) | 14 (16) | 7 (7) | 2 (3) | 1 (1) | 1 (2)
Platelet count decreased (Investigations) | 4 (5) | 7 (7) | 7 (8) | 1 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 7 (8) | 6 (6) | 2 (2) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (4) | 8 (9) | 6 (7) | 1 (2) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (5) | 11 (12) | 11 (11) | 1 (1) | 2 (2) | 1 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 7 (7) | 7 (8) | 1 (3) | 0 (0) | 1 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (5) | 12 (13) | 9 (10) | 2 (4) | 1 (1) | 1 (3)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (4) | 7 (8) | 7 (7) | 1 (1) | 2 (2) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (2) | 9 (9) | 5 (6) | 0 (0) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 3 (4) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (9) | 8 (10) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3) | 8 (8) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Adenocarcinoma (ECF + Cetuximab) (N=67) | Arm B: Adenocarcinoma (IC + Cetuximab) (N=73) | Arm C: Adenocarcinoma (FOLFOX + Cetuximab) (N=73) | Arm A: Squamous Cell Carcinoma (ECF + Cetuximab) (N=8) | Arm B: Squamous Cell Carcinoma (IC + Cetuximab) (N=8) | Arm C: Squamous Cell Carcinoma (FOLFOX + Cetuximab) (N=6)
Blood disorder (Blood and lymphatic system disorders) | 2 (36) | 1 (3) | 2 (21) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 47 (264) | 56 (312) | 49 (326) | 5 (25) | 4 (16) | 4 (35)
Hemolysis (Blood and lymphatic system disorders) | 2 (3) | 4 (10) | 2 (13) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (4) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 2 (15) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 6 (8) | 5 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (2) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 3 (6) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 3 (7) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 14 (30) | 26 (66) | 14 (27) | 2 (3) | 3 (3) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 38 (102) | 39 (94) | 38 (137) | 5 (6) | 2 (3) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 35 (85) | 54 (175) | 45 (162) | 5 (9) | 5 (6) | 4 (9)
Dry mouth (Gastrointestinal disorders) | 4 (11) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 10 (15) | 7 (12) | 11 (23) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 22 (47) | 18 (45) | 14 (51) | 3 (8) | 2 (2) | 1 (4)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 30 (82) | 12 (26) | 18 (54) | 4 (11) | 0 (0) | 2 (13)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 8 (13) | 3 (4) | 2 (3) | 0 (0) | 1 (1) | 1 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (14) | 0 (0) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 4 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 30 (81) | 12 (25) | 29 (94) | 2 (8) | 1 (1) | 2 (8)
Nausea (Gastrointestinal disorders) | 48 (164) | 54 (151) | 42 (175) | 7 (17) | 3 (6) | 5 (16)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (5) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 4 (6) | 7 (12) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (65) | 34 (84) | 33 (61) | 4 (10) | 4 (4) | 4 (10)
Chest pain (General disorders) | 8 (9) | 4 (4) | 7 (23) | 1 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 8 (12) | 12 (21) | 14 (27) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 7 (10) | 14 (24) | 9 (17) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 63 (318) | 65 (330) | 61 (558) | 8 (44) | 6 (8) | 5 (23)
Fever (General disorders) | 4 (6) | 5 (6) | 11 (12) | 0 (0) | 0 (0) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 1 (2) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 12 (19) | 6 (10) | 6 (17) | 0 (0) | 1 (1) | 2 (5)
Visceral edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 8 (9) | 5 (7) | 7 (7) | 0 (0) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 6 (7) | 2 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 5 (7) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 5 (10) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (13)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 5 (6) | 4 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (17) | 23 (47) | 17 (59) | 2 (2) | 1 (1) | 0 (0)
Alkaline phosphatase (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 15 (36) | 24 (62) | 24 (92) | 2 (2) | 2 (7) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 14 (19) | 21 (34) | 27 (91) | 2 (2) | 2 (3) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (2) | 6 (8) | 4 (26) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 18 (57) | 11 (32) | 3 (3) | 2 (4) | 0 (0) | 0 (0)
INR increased (Investigations) | 2 (6) | 2 (3) | 4 (40) | 0 (0) | 2 (2) | 1 (2)
Laboratory test abnormal (Investigations) | 5 (43) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 38 (158) | 39 (165) | 33 (228) | 2 (2) | 2 (10) | 3 (8)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 9 (47) | 13 (54) | 11 (107) | 2 (2) | 1 (5) | 1 (5)
Lymphopenia for pediatric BMT studies (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 51 (228) | 46 (192) | 40 (198) | 7 (33) | 5 (16) | 4 (6)
Platelet count decreased (Investigations) | 25 (74) | 29 (115) | 32 (239) | 3 (14) | 3 (6) | 2 (7)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 4 (10) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 2 (2) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 15 (27) | 24 (53) | 18 (64) | 2 (2) | 3 (12) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 33 (102) | 34 (88) | 35 (130) | 4 (7) | 3 (3) | 2 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 31 (145) | 38 (154) | 31 (225) | 3 (16) | 2 (2) | 3 (24)
Dehydration (Metabolism and nutrition disorders) | 17 (39) | 28 (61) | 14 (34) | 3 (3) | 3 (3) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 18 (59) | 35 (136) | 31 (145) | 1 (13) | 5 (11) | 3 (33)
Serum calcium decreased (Metabolism and nutrition disorders) | 22 (53) | 27 (78) | 18 (69) | 1 (1) | 3 (11) | 3 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (12) | 1 (1) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 7 (11) | 1 (1) | 1 (1) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 40 (180) | 51 (255) | 38 (238) | 5 (34) | 4 (15) | 3 (10)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3) | 5 (9) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 22 (61) | 29 (77) | 31 (91) | 1 (4) | 2 (7) | 3 (10)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (5) | 6 (9) | 7 (13) | 3 (6) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 26 (62) | 34 (79) | 26 (60) | 0 (0) | 3 (7) | 3 (6)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (12) | 5 (18) | 3 (29) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (13) | 12 (22) | 12 (27) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (6) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (8) | 1 (2) | 2 (9) | 0 (0) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (11) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (10) | 6 (11) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (13) | 5 (8) | 7 (51) | 0 (0) | 1 (3) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (7) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 11 (24) | 13 (26) | 13 (18) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 13 (26) | 11 (31) | 19 (111) | 3 (4) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 2 (4) | 5 (9) | 1 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (7) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (5) | 1 (4) | 4 (13) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (117) | 30 (108) | 60 (515) | 6 (14) | 1 (3) | 1 (22)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 2 (9) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (15) | 4 (7) | 7 (31) | 1 (1) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 10 (17) | 5 (7) | 8 (19) | 1 (4) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 10 (22) | 13 (33) | 15 (49) | 0 (0) | 0 (0) | 3 (4)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney pain (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (12) | 1 (1) | 2 (11) | 1 (1) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (18) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (36) | 15 (31) | 15 (45) | 2 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (38) | 20 (49) | 18 (75) | 2 (5) | 0 (0) | 1 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 4 (4) | 11 (40) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 4 (12) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 6 (19) | 2 (3) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 36 (129) | 25 (92) | 24 (117) | 7 (19) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 22 (58) | 16 (40) | 17 (75) | 3 (18) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 21 (53) | 11 (21) | 19 (113) | 3 (9) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 13 (26) | 8 (18) | 12 (63) | 1 (3) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (11) | 6 (11) | 16 (89) | 1 (8) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 42 (201) | 49 (219) | 49 (530) | 5 (35) | 4 (5) | 3 (28)
Rash desquamating (Skin and subcutaneous tissue disorders) | 21 (84) | 16 (59) | 25 (147) | 1 (1) | 0 (0) | 2 (11)
Skin disorder (Skin and subcutaneous tissue disorders) | 7 (11) | 6 (9) | 8 (26) | 1 (7) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 11 (25) | 4 (12) | 0 (0) | 1 (1) | 2 (7)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 5 (5) | 10 (12) | 7 (18) | 1 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less